CLINICAL TRIAL: NCT06871215
Title: Inflammation and Infective Endocarditis
Status: Withdrawn | Type: Observational
Why Stopped: Submission has now been withdrawn
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 19720646
Record Dates: First submitted 2025-01-27; First posted 2025-03-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Infective Endocarditis (IE)
Keywords: Endocarditis; Transcatheter; Valve; Congenital
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells and heart valve tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Native valve: Patients with IE that affects their native heart valve(s).
- Prosthetic valve: Patients with IE that affects an artificial heart valve.
- Cardiac-device related: Patients with IE associated with a cardiac device (e.g. pacemaker).
- Uncorrected congenital: Patients with IE associated with uncorrected congenital heart disease.
- Recurrent: Patients with IE where it is not their first episode

SUMMARY:
Infective endocarditis (IE) is caused by bloodstream bacteria becoming adherent to, and eventually destroying, heart valve tissue. It is a condition that is becoming increasingly common and is associated with significant morbidity and mortality. IE is more common in patients with previous valve replacements and those with congenital heart disease (both corrected and uncorrected). Current treatments in IE are extremely limited; patients are typically managed with intravenous antibiotics and high risk cardiac surgery. Based on unpublished pilot data (valve tissue) from a small cohort of patients (n=3), the investigators hypothesise that the immune system - which is usually responsible for fighting infections - in IE is overactive and may in fact play a role in disease progression. It is possible that adaptive immune cells (B- and T- lymphocytes) that have been exposed to cardiac proteins as a result of bacterial damage, may attack the heart and exacerbate valve destruction. The investigators hypothesise that through the analysis of adaptive immune cells in the blood and valve tissue, it will be possible to identify patients with IE who may have a form of autoimmune heart disease, who might stand to benefit from innovative immune-modulating therapies. To address this hypothesis, the investigators will undertake the following: 1. An observational cohort study in patients with IE to analyse the immune cell status in the peripheral blood and valve tissue (obtained at surgical explant).

DETAILED DESCRIPTION:
Infective endocarditis (IE) is challenging to diagnose despite modern, multi-modality imaging techniques. Its frequency is increasing as more interventions are performed on patients with pre-existing valve disease. Current strategies for diagnosis and management are relatively historical; patients require positive blood cultures and are managed with intravenous antibiotics and cardiac surgery. While the immunological complications of IE are well recognised (e.g. rheumatoid factor positivity), there has been very little research to explore the immune system's role in disease onset and progression. The investigators laboratory has discovered and characterised a group of circulating immune cells (cMET+ T-cells) that appear to have a direct role in the progression of another inflammatory heart disease known as myocarditis. Pilot data from the investigators laboratory (n=3 patients) suggests that these cells are also detectable in explanted valve tissue from patients undergoing endocarditis surgery. The investigators suspect that the presence of these cells in IE implies that there may be a significant contribution to disease progression from the immune system. It is possible that the exposure of cardiac proteins by damage caused by a bacterial infection primes the immune system against self, and that these auto-reactive T-cells then go on to attack and destroy native valve tissue. The investigators would like to investigate whether circulating and myocardial cMET+ T-cells are detectable across the wide spectrum of patients with IE and further explore their role in this condition. The investigators are planning to functionally characterise both circulating cells and those that are detectable in explanted valve tissue using a combination of flow cytometry and spatial RNA sequencing. The investigators propose that cMET+ T-cells may have utility in the diagnosis of IE and that in patients with a significantly elevated number, the investigators might be able to offer novel (and highly specific) targeted immunological therapy that could improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of infective endocarditis according to the Duke Criteria.

Exclusion Criteria:

* Active solid organ or haematological malignancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 100 patients with infective endocarditis who will be recruited from within Barts Health NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral and valvular cMET+ T-cell frequency | 18 months
  The proportion of T-cells in the peripheral blood and myocardial valve tissue that express the receptor cMET, which has been described as a marker of cardiac autoimmunity will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Peripheral and valvular T-cell phenotype | 18 months
  Pre-defined T-cell flow cytometry panels will be used to interrogate the expression of various surface and intracellular markers (activation, memory status, cytokine expression) on peripheral and valvular T-cells.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Marelli-Berg, MD PhD, Study Director — Queen Mary University of London; Simon Woldman, MD, Study Director — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT06871215/Prot_000.pdf
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT06871215/ICF_001.pdf